CLINICAL TRIAL: NCT03191058
Title: Confirmatory Efficacy and Safety Trial of Magnetic Seizure Therapy for Depression (CREST - MST)
Brief Title: Confirmatory Efficacy and Safety Trial of Magnetic Seizure Therapy for Depression
Acronym: CREST-MST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Centre for Addiction and Mental Health (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Carol A. Tamminga, Professor and Chairperson, Department of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 032017-022; 1R01MH112815-01 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Depression; Unipolar Depression; Treatment Resistant Depression
Keywords: Depression; Unipolar Depression; Treatment Resistant Depression; Magnetic Seizure Therapy; Suicidal Ideation; Electroconvulsive Therapy
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double blind, parallel--group clinical trial with two treatment arms conducted both at the University of Texas Southwestern in Dallas, Texas and at the Temerty Centre for Therapeutic Brain Intervention based at CAMH in Toronto, Canada. Both sites aim to recruit 130 participants each.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomized into the study using a permuted block method with a random number generator. The study statistician will prepare the randomization scheme. The block size will be varying and study personnel will be blinded to the randomization block size.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Magnetic Seizure Therapy (MST) (Experimental): MST treatments will be administered using the MagPro MST with Cool TwinCoil.
  Interventions: Device: Magnetic Seizure Therapy
- Electroconvulsive Therapy (ECT) (Active Comparator): ECT treatments will be administered using the MECTA spECTrum 5000Q or the MECTA Sigma devices.
  Interventions: Device: Electroconvulsive Therapy

INTERVENTIONS:
Device: Magnetic Seizure Therapy — MST treatment will be administered using the MagPro MST with a Cool TwinCoil over the frontal cortex in the midline position using 100 Hz stimulation. The MST determination of seizure threshold will be done using 100% machine output applied at 100 Hz at progressively escalating train durations, commencing at 2 seconds and increasing by 2 seconds with each subsequent stimulation until an adequate seizure is produced. During subsequent sessions, one stimulation will be delivered using a train duration that is 4 seconds longer than the train duration at threshold (with a maximum train duration of 10 seconds).
  This will be performed under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes.
  Other Names: MST
  Arms: Magnetic Seizure Therapy (MST)
Device: Electroconvulsive Therapy — In the ECT arm treatment, the MECTA spectrum 5000Q or the MECTA Sigma devices will be used, which are FDA approved devices used for providing standard-of-care clinical ECT treatments. The ECT determination of seizure threshold and the adjustment of energy at subsequent sessions will be based on a standard published protocol. All participants will receive RUL-UB ECT at six times the seizure threshold under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes
  Other Names: ECT
  Arms: Electroconvulsive Therapy (ECT)

SUMMARY:
This trial aims to assess the efficacy and tolerability of Magnetic Seizure Therapy (MST) as an alternative to electroconvulsive therapy (ECT) for depression. Even with multiple medication trials, 30 - 40% of patients will experience a pharmacologically resistant form of illness. The ineffectiveness of current treatments for major depressive disorder (MDD) coupled with the economic burden associated with the disorder engenders a need for novel therapeutic interventions that can provide greater response and remission rates.

DETAILED DESCRIPTION:
The study will involve a randomized, double blind, non-inferiority clinical trial with two treatment arms conducted in two international academic medical centers (the Centre for Addiction and Mental Health in Toronto, Canada and UT Southwestern in Dallas, Texas). The investigators are pursuing a non-inferiority clinical trial in an effort to compare MST - a new treatment for TRD - to RUL-UB-ECT. Treatment will be administered two to three days per week. Depression symptoms will be assessed with the 24-item Hamilton Depression Rating Scale (HRSD-24) and suicidality will be assessed with the Scale for Suicidal Ideation (SSI). Remission will be defined as HRSD-24 < or = 10 and a > 60% decrease in scores from baseline on two consecutive ratings. Once a participant reaches remission, a second rating to confirm remission will be conducted immediately before their next scheduled treatment. If remission is confirmed, they will then be considered a completer of the acute treatment course. Remission of suicidal ideation is defined as a score of 0 on the SSI. Therefore, there will be no specific minimum number of treatments that patients must receive to be classified as remitters. However, patients who do not meet remission criteria after 21 treatment sessions will be considered non-remitters and will cease treatment sessions. This maximum treatment number was chosen allowing for the possibility that MST may require more treatment sessions to achieve remission, similar to RUL-UB ECT. The blind will not be broken to participants until the completion of the entire study.

ELIGIBILITY:
Inclusion Criteria

Patients will be included if they:

1. are inpatients or outpatients;
2. are voluntary and competent to consent to treatment and research procedures according to ECT/MST attending psychiatrist;
3. have a MINI International Neuropsychiatric Interview diagnosis, Version 6 (MINI-6.0) diagnosis of non-psychotic MDD
4. are 18 years of age or older
5. have a baseline HRSD-24 score > or = 21;
6. are considered to be appropriate to receive convulsive therapy as assessed by an ECT attending psychiatrist and a consultant anaesthesiologist
7. are agreeable to keeping their current antidepressant treatment constant during the intervention;
8. are likely able to adhere to the intervention schedule;
9. meet the MST safety criteria [75];
10. If a woman of child-bearing potential: is willing to provide a negative pregnancy test and agrees not to become pregnant during trial participation.

Exclusion Criteria

Patients will be excluded if they:

1. have a history of MINI diagnosis of substance dependence or abuse within the past three months;
2. have a concomitant major unstable medical illness;
3. are pregnant or intend to get pregnant during the study;
4. have a MINI diagnosis of any primary psychotic disorder
5. have a MINI diagnosis of obsessive compulsive disorder, or post-traumatic stress disorder deemed to be primary and causing more functional impairment than the depressive disorder
6. have probable dementia based on study investigator assessment;
7. have any significant neurological disorder or condition likely to be associated with increased intracranial pressure or a space occupying brain lesion, e.g., cerebral aneurysm;
8. present with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, rheumatoid arthritis requiring high dose prednisone, or Cushing's disease);
9. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
10. require a benzodiazepine with a dose > lorazepam 2 mg/day or equivalent or any anticonvulsant due to the potential of these medications to limit the efficacy of both MST and ECT;
11. are unable to communicate in English fluently enough to complete the neuropsychological tests;
12. have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Improvement in symptom severity of depression as measured by the Hamilton Rating Scale for Depression - 24 (HRSD-24) | 7 weeks
  Hamilton Rating Scale for Depression (24-item version):
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-76 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Cognitive adverse effects as indexed by the Autobiographical Memory Test (AMT) | 7 weeks
  Autobiographical Memory Test:
  -Interviewer-rated measure with 10 items that indexes autobiographical memory recall and specificity.

SECONDARY OUTCOMES:
Improvement in symptom severity of Suicidal Ideation as measured by the Scale for Suicidal Ideation (SSI) | 7 weeks
  Scale for Suicidal Ideation:
  * This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas
  * Scale range: 0 - 38 (total score)
  * Lower scores indicate lower severity of suicidal ideation (i.e., better outcome)
  * Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (3):
- United States (2):
  - University of California San Diego, San Diego, California
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daskalakis ZJ, McClintock SM, Hadas I, Kallioniemi E, Zomorrodi R, Throop A, Palmer L, Farzan F, Thorpe KE, Tamminga C, Blumberger DM. Confirmatory Efficacy and Safety Trial of Magnetic Seizure Therapy for Depression (CREST-MST): protocol for identification of novel biomarkers via neurophysiology. Trials. 2021 Dec 11;22(1):906. doi: 10.1186/s13063-021-05873-7. PMID 34895296
- [Derived] Daskalakis ZJ, Tamminga C, Throop A, Palmer L, Dimitrova J, Farzan F, Thorpe KE, McClintock SM, Blumberger DM. Confirmatory Efficacy and Safety Trial of Magnetic Seizure Therapy for Depression (CREST-MST): study protocol for a randomized non-inferiority trial of magnetic seizure therapy versus electroconvulsive therapy. Trials. 2021 Nov 8;22(1):786. doi: 10.1186/s13063-021-05730-7. PMID 34749782
- [Derived] Regenold WT, Deng ZD, Lisanby SH. Noninvasive neuromodulation of the prefrontal cortex in mental health disorders. Neuropsychopharmacology. 2022 Jan;47(1):361-372. doi: 10.1038/s41386-021-01094-3. Epub 2021 Jul 16. PMID 34272471
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914